CLINICAL TRIAL: NCT03119857
Title: A Randomized, Open Label, Multicenter, Phase III, 2-Arm Study of Androgen Deprivation +/- Taxotere (Docetaxel) for Non-metastatic Prostate Cancer Patients With a Rising PSA
Brief Title: Early Rising PSA Endocrine Treatment Versus Chemo-endocrine Therapy- SPCG14
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Josefsson, PI, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 1.6
Record Dates: First submitted 2016-05-14; First posted 2017-04-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Prostatic Neoplasms
Keywords: Non-metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiandrogen (Active Comparator): Antiandrogen (bicalutamide 150 mg x 1) p.o. alone,
  Interventions: Drug: Antiandrogen
- Antiandrogen + docetaxel (Experimental): Antiandrogen (bicalutamide 150 mg x 1) p.o. + Docetaxel 75 mg/m2 (maximum 2.0 m2 ) i.v. q 3 weeks x up to 8-10 cycles.
  Interventions: Drug: Antiandrogen+docetaxel

INTERVENTIONS:
Drug: Antiandrogen
  Arms: Antiandrogen
Drug: Antiandrogen+docetaxel — Antiandrogen (bicalutamide 150 mg x 1) + docetaxel (Taxotere®) 75mg/m2 (max 2.0m2) i.v. in 60 minutes on day 1. One cycle is 21 days. Docetaxel will be given for up to 8-10 cycles or until unacceptable toxicity or consent withdrawal whichever comes first.
  Antiemetic therapy may be used if necessary.
  Other Names: Taxotere
  Arms: Antiandrogen + docetaxel

SUMMARY:
Summary

In patients with prostate cancer (PC) who have only biochemically relapsed disease after curative treatment (or some locally advanced PC patients), hormonal therapy remains a de facto standard of care treatment. Adding docetaxel-based chemotherapy to a standard-of-care hormonal therapy has an increased potential to treat prostate cancer cell clones resistant to androgen withdrawal and to possibly shorten the duration of therapy needed to control the disease.

This clinical trial is designed on the basis of an unmet clinical need, as well as other factors including: 1) a consensus among investigators on endpoints for studies of patients with a rising PSA, 2) the ability to identify subjects at high risk for developing radiographic metastases, 3) the fact that hormonal therapy has already been shown to improve survival when applied early in the natural history, and 4) the availability of chemotherapy such as docetaxel that can improve survival in subjects with advanced disease.

It is our hypothesis that a more appropriate group of patients who may benefit from the curative potential of systemic chemo-hormonal modality is that with minimal, but detectable disease who have a high probability of developing metastatic disease, clinical symptoms and eventually death from prostate cancer in a defined time frame. The investigators hypothesize further that the approach is likely to be more effective at a time of minimal tumour burden, resulting in minimization of the overall burden of therapy and better quality of life while on treatment.

This trial will determine whether any benefit is gained by adding chemotherapy to hormonal therapy alone in the population of subjects with a rising PSA. Two therapeutic approaches will be compared in this two-arm randomized clinical trial. The control Arm A provides antiandrogen (bicalutamide 150 mg x 1) alone. The experimental Arm B involves treatment with docetaxel for 8-10 cycles and antiandrogen (bicalutamide 150 mg x 1) treatment. For the schematic representation of study design please see Section 7.3.1.

Subjects with a rising PSA following definitive local curative therapy will be eligible, if their PSA doubling time is < 12 months. Also PC patients planned for anti-.androgen therapy are eligible, with the same criteria. Subjects with radiographic metastases will be excluded. The primary endpoint of the trial is progression-free survival of subjects that do not experience biochemical failure at 60 months from the start of therapy.

Based on the yearly number of prostate cancer patients who undergo definitive local therapies and the estimated probabilities of relapse, upwards of 400 men (if +15% improvement) in the Scandinavian countries are potential candidates for this approach.

ELIGIBILITY:
Inclusion Criteria:

* Men > 18 and ≤80 years of age.
* WHO/ECOG performance status 0 - 1 (WHO: World Health Organization; ECOG: Eastern Cooperative Oncology Group )
* Histological proven adenocarcinoma of the prostate.
* Patients who are planned to receive antiandrogen (bicalutamide 150 mg x 1) treatment,
* After curative treatment

  * Prostatectomy: PSA > 10 OR PSA DT < 12 months and PSA > 0.5 (PSA doubling time calculation must start at a minimum value of > 0.5)
  * Radiation: PSA > +2.0 above nadir and PSA >10 OR PSA DT < 12 months and PSA > 0.5. (PSA bouncing after radiotherapy should be excluded according to the local traditions, and PSA doubling time calculation must start at a minimum value of > 0.5)
* In locally advanced (or local not suitable for curative therapy) prostate cancer patients, PSA < 100 is required before inclusion AND one of the following

  * PSA DT < 12 months or
  * PSA >20 or
  * Gleason score 8-10
* Previous hormonal therapy in conjunction with radiotherapy is allowed, provided that the total duration of therapy does not exceed 12 months and has to be stopped > 12 months ago.
* Testosterone value > 5 nmol/l
* Adequate haematological-, liver- and kidney function. WBC(white blood cell ) 3.5 x 109/L ANC(absolute neutrophil count ) 1.5 x 109/L Platelet Count 150 x 109/L Haemoglobin > 120 g/L Total bilirubin ≤ ULN (upper limit of normal) unless due to Gilbert's disease Creatinine ≤ 1.5 x ULN or creatinine clearance of 60 cc/min or corresponding Iohexol clearance value ASAT(aspartate aminotransferase )/ALAT(alanine aminotransferase) ≤ 1.5 x ULN ALP (Alkaline phosphatase) < 1.5 x ULN
* Negative bone scan performed no more than 3 months prior to randomisation.
* Additional CT or ultrasound of thorax, abdomen and/or pelvis is optional.
* Written informed consent.

Exclusion Criteria:

* Positive bone scan
* Any distant metastasis detected by CT or ultrasound
* Patients with a history of previous malignant disease. Exceptions should be made for basal cell carcinoma (BCC) and squamous cell carcinoma of the skin. Exceptions should also be made for curatively treated malignant disease, which has been disease free for the past 5 years.
* Previous chemotherapy or randomised in SPCG 12/AdPro or SPCG 13/AdRad (SPCG: Scandinavian Prostate Cancer Group).
* Systemic corticosteroids within 6 months prior to randomisation.
* Unstable cardiovascular disease, including myocardial infarction, within 6 months prior to randomisation.
* Active untreated infectious disease, including tuberculosis, MRSA (Methicillin-resistant Staphylococcus aureus.
* Active gastric ulcer.
* Known hypersensitivity to Polysorbate 80 (an excipient of docetaxel)
* Other serious illness or medical condition
* Symptomatic peripheral neuropathy ≥ CTCAE grade 2.
* Patients who by altered physical or psychological state not are able to co-operate or participate in the trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, which ever came first, assessed up to 60 months
  Progression free survival defined as the time from randomization to the date of first documentation of:
  * PSA progression PSA progression is considered to occur when PSA is +2.0 ng/ml above nadir. A confirmatory PSA must be taken no less than 6 weeks following the first rising PSA above nadir +2.0 ng/ml. If that confirmatory PSA also exceeds the above parameters, then progression has occurred. If the confirmatory PSA fails to confirm progression, then the patient will remain on study.
  * Radiographic progression Outcome in patients who develop radiographically metastatic disease while on study will be defined as progression independent of their respective PSA values.
  These patients will be followed for evaluation of survival.
  - Death Death due to prostate cancer in the absence of previous documentation of disease progression,

SECONDARY OUTCOMES:
Difference between groups in PSA doubling time (PSADT). | From date of randomization until the date of first documented PSADT, assessed up to 60 months
  The PSADT can be calculated by the natural log of 2 (0.693) divided by the slope of the relation between the log of PSA and the time of PSA measurement.
Difference between groups regarding QoL | At date of randomization and yearly, assessed up to 60 months
  The quality of life (QoL) will be assessed using the FACT-P-T disease-specific subscale. The scoring will be in accordance with version 4 of the FACT manual.
Difference between groups regarding metastasis free survival | From date of randomization until the date of first documented date of metastases, assessed yearly by bone-scan after first PSA_progression until first sign of metastasis, whichever came first, assessed up to 100 months
  Metastasis free survival will be assessed yearly by bone-scan after first PSA progression until the date of first documented metastasis on bone scan, date of death from any cause, whichever came first, assessed up to 100 months
Difference between groups regarding overall survival | From date of randomization until the date of death from any cause reported yearly by the study sites up to 100 months
  Survival will be assessed yearly up to 100 months after inclusion
Difference between groups regarding cancer specific survival | From date of randomization until date of death from prostate cancer,reported yearly by the study sites up to 100 months
  Cancer specific survival will be assessed yearly up to 100 months after inclusion
Measurement of grade of toxicity of given treatments | At date of randomization, during treatment and follow up questionaries until 60 months
  Adverse events recording using NCI-CTCAE (v3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Josefsson, PhD, Principal Investigator — Univeristy of Gothenburg; Ingela Turesson, Prof, Principal Investigator — Uppsala University
Locations (5):
- Copenhagen University hospital, Rigshospitalet, Copenhagen, Denmark
- Finland (2):
  - Kuopio University Hospital, Kuopio, Kuopio Kuopio
  - Turku University Hospital, Turku
- Erasmus Medical Center Rotterdam, Rotterdam, Netherlands
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- See also: SPCG home — http://spcg.se/trials/spcg-14-spcg-14-psa-erect-m0/